CLINICAL TRIAL: NCT01021605
Title: A Prospective, Non-Randomized Feasibility Study of the Hemolung Respiratory Assist System in Patients With Acute Hypercapnic Respiratory Failure
Brief Title: Feasibility Study of the Hemolung Respiratory Assist System (Germany)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alung Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-CA-1000
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Hypercapnic Respiratory Failure, COPD, ARDS
Keywords: hypercapnic respiratory failure, COPD, ARDS
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemolung Respiratory Assist System (Experimental)
  Interventions: Device: Hemolung Respiratory Assist System

INTERVENTIONS:
Device: Hemolung Respiratory Assist System — Patients meeting the inclusion criteria will be placed on the Hemolung Respiratory Assist System. Patients will be weaned from non-invasive or invasive ventilation and then the Hemolung RAS. Hemolung support will be provided for up to 7 days. Follow-up exams will be performed every 15 days until hospital discharge or 30 days from completion of Hemolung therapy, whichever is later.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Hemolung Respiratory Assist System (RAS) in patients with hypercapnic respiratory failure.

DETAILED DESCRIPTION:
The objective of the feasibility study is to evaluate the safety and efficacy of the Hemolung RAS in patients with hypercapnic respiratory failure in five groups of patients:

Group 1: COPD patients with an acute exacerbation and have a 50% likelihood of failure of noninvasive positive pressure ventilation (NIPPV) leading to intubation and mechanical ventilation

Group 2: Patients with hypercapnic respiratory failure on invasive mechanical ventilation who have either:

* Failed two or more weaning attempts OR
* Failed one or more weaning attempts and do not wish to be invasively mechanically ventilated.

Group 3: Patients with hypercapnic respiratory failure on noninvasive positive pressure ventilation who have failed two weaning attempts and do not wish to be invasively mechanically ventilated.

Group 4: Patients with hypercapnic respiratory failure who in the view of the treating physician are declining on optimized non-invasive positive pressure ventilation OR demonstrate a complete intolerance of non-invasive positive pressure ventilation for any reason and invasive mechanical ventilation is considered undesirable by the treating physician.

Group 5: Patients who are currently invasively mechanically ventilated and in the view of the treating physician would benefit from the application of protective lung ventilation, and in whom this cannot be achieved without significant worsening of respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed hypercapnic respiratory failure (PaCO2 >50mmHg(6.7kPa)) and falling into one of the five groups
* Not severely hypoxemic (PaO2/FiO2 ≥ 200 mmHg on PEEP/CPAP ≤ 5 cmH2O)
* Hemodynamically stable: Mean arterial pressure (MAP) > 65 mmHg without vasopressor support, or MAP > 60 mmHg with a requirement for vasopressor support that can be attributed to sedation or dynamic hyperinflation resulting from mechanical ventilation by the treating investigator.
* Chronic arrhythmias (e.g., atrial fibrillation) well controlled
* Minimum platelet count of 100,000/mm3
* Minimum red blood cell count of 2.5 mill/μl

Group 1:

* Known or suspected severe COPD, as defined by the GOLD criteria
* On non-invasive positive pressure mechanical ventilation > 1hour with either:
* PaCO2 > 55 mmHg with pH < 7.25 OR
* PaCO2 > 55 mmHg with < 5mmHg decrease from baseline and pH < 7.30

Group 2:

* Intubated or tracheostomized patients with hypercapnic respiratory failure who either:
* Has failed at least 2 weaning attempts or
* Has failed at least 1 attempt and wishes not to be invasively mechanically ventilated

Group 3:

* Patient on NIPPV due to hypercapnic respiratory failure who has failed at least 2 weaning attempts and has refused intubation

Group 4:

* Patients with hypercapnic respiratory failure who are failing optimal NIPPV or demonstrate a complete intolerance to NIPPV and IMV is considered undesirable

Group 5:

* Patients who are on IMV and would benefit from the application of lung protective ventilation, and in whom this would not be achieved without significant worsening of respiratory failure
* On IMV for at least 12 hours
* pH <7.30 due to respiratory acidosis

Exclusion Criteria:

* Presence of acute, uncontrolled arrhythmia
* Acute ischemic heart disease
* Presence of bleeding diathesis
* Significant abnormality or weakness/paralysis of respiratory muscles due to a know muscular dystrophy or neurologic disorder
* Recent (< 7 days) prolonged (>24 hrs) use of muscle paralyzing agents
* Cerebrovascular accident, intracranial bleed, head injury or other neurologic disorder likely to affect ventilation
* Coma from any cause, or decreased consciousness
* Hypersensitivity to heparin or previous heparin induced thrombocytopenia
* Recent (< 6 months) major chest abdominal trauma or surgery
* Presence of septic shock
* Presence of a significant pneumothorax or bronchopleural fistula
* History of uncontrolled major psychiatric disorder
* Pregnant women
* Known to have AIDS or to have symptomatic HIV
* Received chemotherapy or radiation within the previous 90 days
* Received an organ transplant other than corneal transplants
* Received or currently receiving immunosuppressive therapy, excluding corticosteroids within the last 3 months
* Presence of severe renal or liver failures
* Known vascular abnormality which would complicate or prevent successful insertion of the vascular access catheter in either the right internal jugular vein or right femoral vein
* Presence of another catheter in both the right internal jugular vein and right femoral vein that cannot be moved to allow insertion of the Hemolung catheter in one of these vessels.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The ability of the Hemolung to remove a minimum of 50 mL/min of CO2 for up to seven days and reliable performance of the device over the length of use | 7 days
The frequency of occurrence of serious adverse events while on Hemolung therapy and up to 30 days from completion of Hemolung therapy. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Felix JF Herth, MD, Principal Investigator — Thoraxklinik-Heidelberg gGmbH
Locations (7):
- Germany (7):
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Ruhrlandklinik Das Lungenzentrum Essen-Heidhausen Abt.: Pneumologie, Essen, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Bonn
  - Klinik Donaustauf, Donaustauf
  - Universitätsmedizin Göttingen, Göttingen
  - Asklepios Klinik Barmbek, Hamburg
  - Krankenhaus Bethanien, Solingen

REFERENCES:
- [Derived] Burki NK, Mani RK, Herth FJF, Schmidt W, Teschler H, Bonin F, Becker H, Randerath WJ, Stieglitz S, Hagmeyer L, Priegnitz C, Pfeifer M, Blaas SH, Putensen C, Theuerkauf N, Quintel M, Moerer O. A novel extracorporeal CO(2) removal system: results of a pilot study of hypercapnic respiratory failure in patients with COPD. Chest. 2013 Mar;143(3):678-686. doi: 10.1378/chest.12-0228. PMID 23460154